CLINICAL TRIAL: NCT05788042
Title: Randomised Controlled Trial of Neurostimulation for Symptoms of Anorexia Nervosa
Brief Title: Trial of Enhanced Neurostimulation for Anorexia
Acronym: TRENA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-016
Record Dates: First submitted 2023-02-21; First posted 2023-03-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-04

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Repetitive Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation; Non-invasive brain stimulation
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, sham-controlled trial, parallel group design. Participants will be randomised to one of four groups (2:1:2:1 ratio): Active or sham tDCS, or Active or sham rTMS. The brain stimulation protocols involve 84 sessions of tDCS (active or sham) or 56 sessions of rTMS (active or sham) over the 8 week acute treatment period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial participants, their treating psychiatrist, ward staff, and a study staff member (who will conduct blinded assessments of mood secondary outcome measures) will be blinded after assignment to intervention until the database is locked and the primary analysis completed. The following measures will be taken to ensure preservation of blinding to treatment allocation:
  * Unblinded personnel (i.e., Neurostimulation Nurse(s) and/or tDCS research assistant), will be present during rTMS treatment delivery. tDCS will be self administered in the presence of ward staff. Team members involved in conducting blinded assessments for mood (i.e., MADRS) must not be present in the room during research treatment delivery.
  * Knowledge of the code (i.e., which of 'A', 'B', 'C' or 'D' refers to which randomised treatment) will only be known to study staff responsible for treatment delivery, the study CI and study statistician involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active transcranial Direct Current Stimulation (tDCS) (Active Comparator): It will be given continuously for 30 minutes at 2 mA, twice daily (separated by >=2 hours) over the first 4 weeks, and daily over the second 4 weeks of the 8 week acute treatment period (84 sessions total).
  Interventions: Device: tDCS mini-CT Stimulator (Soterix, USA: ARTG: 284637)
- Sham transcranial Direct Current Stimulation (tDCS) (Sham Comparator): It will involve an initial ramping up to 0.5 mA and then a ramp down to 0 mA for the remainder of each treatment. The same number of sessions as active tDCS will be administered.
  Interventions: Device: tDCS mini-CT Stimulator (Soterix, USA: ARTG: 284637)
- Active Repetitive Transcranial Magnetic Stimulation (rTMS) (Active Comparator): Active rTMS twice per day (separated by ≥ 2 hours) over the first 4 weeks. Two sessions per day (separated by ≥ 2 hours), given on 2 days each week for the following 4 weeks. The total number of rTMS sessions over the 8 week acute treatment period will be 56.
  Interventions: Device: MagPro TMS device (ARTG: 204659)
- Sham Repetitive Transcranial Magnetic Stimulation (rTMS) (Sham Comparator): Sham rTMS twice per day (separated by ≥ 2 hours) over the first 4 weeks. Two sessions per day (separated by ≥ 2 hours), given on 2 days each week for the following 4 weeks. The same number of sessions as active rTMS will be administered.
  Interventions: Device: MagPro TMS device (ARTG: 204659)

INTERVENTIONS:
Device: MagPro TMS device (ARTG: 204659) — rTMS will be administered using a MagPro TMS device (ARTG: 204659) which is approved for its intended use in this trial. rTMS involves the application of transient magnetic pulses which induce small currents in the underlying cortex via the principal of electromagnetic induction. rTMS will be administered using a patterned frequency stimulus called intermittent theta-burst stimulation (iTBS).This form of rTMS was chosen because a recent large multicentre trial showed 3 minutes of iTBS attained the same therapeutic effect as 30 minutes of standard rTMS, leading to FDA approval for depression. Each treatment session will comprise an extended iTBS session, i.e., 6.6 mins, delivered at 100% resting motor threshold (RMT). It will be targeted to the left DLPFC (F3 using the 10-20 International EEG system), consistent with the prior RCT of rTMS for AN.
  Arms: Active Repetitive Transcranial Magnetic Stimulation (rTMS); Sham Repetitive Transcranial Magnetic Stimulation (rTMS)
Device: tDCS mini-CT Stimulator (Soterix, USA: ARTG: 284637) — tDCS will be self-administered using the 1x1 tDCS mini-CT Stimulator (Soterix, USA: ARTG: 284637) with two saline-soaked sponge electrodes held in place on the scalp using the Soterix Ole-2 headband. The device is intended to treat different neurological and psychiatric disorders. tDCS involves the passing of weak electrical current through the brain via electrodes placed upon the scalp. The current modulates the resting membrane potential of stimulated neurons which causes changes in neuronal excitability. The anode will be placed over the left F3 (10-20 System) and the cathode over F4 (electrode sizes 5 x 5cm, 25cm2). This montage was chosen to target the left DLPFC, consistent with prior pilot studies of tDCS in AN.
  Arms: Active transcranial Direct Current Stimulation (tDCS); Sham transcranial Direct Current Stimulation (tDCS)

SUMMARY:
Preliminary open-label studies have suggested that non-invasive brain stimulation methods of both transcranial direct current stimulation (tDCS) and repetitive transcranial magnetic stimulation (rTMS) have clinical benefits for improving psychological and eating disorder related symptoms, which can persist at long-term follow ups after acute treatment (i.e., at 6 and 12 months).

Here the investigators propose to conduct the first double-blinded, randomised sham-controlled study to directly compare the therapeutic effectiveness and acceptability of both treatment modalities.

Participants will be recruited and treated at one inpatient setting (Northside Clinic, St Leonards, Sydney). This facility is one of the largest specialist eating disorder settings in Australia with approximately 130 new admissions every year (2019 data). All participants who give consent and who fulfill the eligibility criteria will be randomised to receive active tDCS, sham (placebo) tDCS, active rTMS or sham rTMS over 8 weeks. Trial participants, their treating psychiatrist, ward staff, and a study staff member (who will conduct blinded assessments of mood secondary outcome measures) will be blinded after assignment to intervention until the database is locked and the primary analysis completed. All participants will complete assessments of eating disorder symptoms, mood, psychological symptoms, neurocognition and functioning at baseline, end of week 4, 8 and 20.

Expected outcomes include data on the relative effectiveness and acceptability for both treatment modalities in the inpatient and at-home setting (i.e., for at-home tDCS). The investigators expect that both active treatment arms will produce clinical benefits and have high acceptability, and that clinical benefits will be maintained with long-term at-home tDCS continuation treatment. These outcomes have potential to assist in reducing hospital stay and emergency re-admissions and improving day to day functioning in participants. Health economic data for both treatment modalities will additionally have utility from a service perspective, given the disparity in resource requirements between the two treatments (TMS, tDCS) in terms of costs for patients and access to treatment for people living in remote and rural areas (i.e., for at-home tDCS).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥16 years,
* A current Diagnostic and Statistical Manual of Mental Disorders (5th edition DSM-5) diagnosis of anorexia nervosa
* Willing and able to participate and comply with study requirements
* Worked or studied in a context requiring some proficiency in spoken English (to ensure validity of neuropsychological testing)
* Under ongoing care by his/her own treating psychiatrist (to ensure patient safety during the study)

Exclusion Criteria:

* Inability to provide informed consent
* Contraindications to tDCS/rTMS
* Failed to respond to an adequate course or rTMS (4 weeks) within the current illness course
* Had ECT in the last 3 months
* MoCA score of <26
* Significant risk of significant self harm or suicide as assessed by study psychiatrist(s)
* Currently enrolled in another interventional clinical trial or using an investigational device/product

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness - Eating Disorder Examination Questionnaire (EDE Q) | Change from baseline at 8 weeks
  Self-report instrument that measures eating disorder behaviors and attitudes. Eating Disorder Examination Questionnaire; 28-items; rating scale 0 - 6; Higher scores on the global scale and subscales indicate more problematic eating behaviours and attitudes.
Acceptability | 8 weeks
  Number of completed sessions for active tDCS and active rTMS in the acute 8 week RCT period.

SECONDARY OUTCOMES:
Weight | Change from baseline at 4 weeks
  Change in Body Mass Index. Weight status in AN is considered a key determinant of remission from illness.
Weight | Change from baseline at 8 weeks
  Change in Body Mass Index. Weight status in AN is considered a key determinant of remission from illness.
Weight | Change from baseline at 20 weeks
  Change in Body Mass Index. Weight status in AN is considered a key determinant of remission from illness.
Mood - Montgomery Asberg Depression Rating Score (MADRS) | Change from baseline at 4 weeks
  Depressive symptomology is a common psychiatric comorbidity of AN and both tDCS and rTMS significantly improve mood symptoms. 10-items; rating scale 0- 6; Higher score indicates more severe depression.
Mood - Montgomery Asberg Depression Rating Score (MADRS) | Change from baseline at 8 weeks
  Depressive symptomology is a common psychiatric comorbidity of AN and both tDCS and rTMS significantly improve mood symptoms. 10-items; rating scale 0- 6; Higher score indicates more severe depression.
Mood - Montgomery Asberg Depression Rating Score (MADRS) | Change from baseline at 20 weeks
  Depressive symptomology is a common psychiatric comorbidity of AN and both tDCS and rTMS significantly improve mood symptoms. 10-items; rating scale 0- 6; Higher score indicates more severe depression.
Neurocognition - Trail Making Test parts A and B (TMT: attention and cognitive flexibility) | Change from baseline at 8 weeks
  Deficits in set shifting has been found to be common in people with AN.
Neurocognition - Trail Making Test parts A and B (TMT: attention and cognitive flexibility) | Change from baseline at 20 weeks
  Deficits in set shifting has been found to be common in people with AN.
Neurocognition - Embedded Figures Test (EFT: field dependence vs independence). | Change from baseline at 8 weeks
  This task assesses central coherence, or the degree of focus on details in processing information. Poor central coherence is a potential etiologic or maintaining factor for people with eating disorders.
Neurocognition - Embedded Figures Test (EFT: field dependence vs independence). | Change from baseline at 20 weeks
  This task assesses central coherence, or the degree of focus on details in processing information. Poor central coherence is a potential etiologic or maintaining factor for people with eating disorders.
Neurocognition - STROOP Colour Word Test (response inhibition). | Change from baseline at 8 weeks
  The STROOP task assesses inhibitory control, which has been shown to be reduced in people with eating disorders.
Neurocognition - STROOP Colour Word Test (response inhibition). | Change from baseline at 20 weeks
  The STROOP task assesses inhibitory control, which has been shown to be reduced in people with eating disorders.
Neurocognition - Wisconsin Card Sorting Test (WSCT: perseveration). | Change from baseline at 8 weeks
  This task has been found to be sensitive to set shifting deficits in people with AN.
Neurocognition - Wisconsin Card Sorting Test (WSCT: perseveration). | Change from baseline at 20 weeks
  This task has been found to be sensitive to set shifting deficits in people with AN.
Psychological Symptoms - Depression Anxiety and Stress Scale (DASS-21) | Change from baseline at 8 weeks
  Self reported questionnaire designed to measure the severity of a range of symptoms common to both Depression and Anxiety. 21-items; rating scale 0- 3; Higher scores on subscales indicate more severe depression, anxiety and stress.
Psychological Symptoms - Depression Anxiety and Stress Scale (DASS-21) | Change from baseline at 20 weeks
  Self reported questionnaire designed to measure the severity of a range of symptoms common to both Depression and Anxiety. 21-items; rating scale 0- 3; Higher scores on subscales indicate more severe depression, anxiety and stress.
Functioning - The Assessment of Quality of Life Instrument (AQoL-4D) | Change from baseline at 8 weeks
  Measures quality of life for independent living, mental health, relationships, and senses. It as chosen as measures can be used for economic evaluation based on Quality Adjusted Life Years (QALYs). 12-items; scale 1-4; Higher score indicates lower health-related quality of life.
Functioning - The Assessment of Quality of Life Instrument (AQoL-4D) | Change from baseline at 20 weeks
  Measures quality of life for independent living, mental health, relationships, and senses. It as chosen as measures can be used for economic evaluation based on Quality Adjusted Life Years (QALYs). 12-items; scale 1-4; Higher score indicates lower health-related quality of life.
Change in Circumplex Scales of Interpersonal Efficacy (CSIE-32) | Change from baseline at 8 weeks
  Change in Circumplex Scales of Interpersonal Efficacy: 32-items; scale 0-10; Higher score indicate confidence that one can engage in variety of interpersonal behaviours.
Change in Circumplex Scales of Interpersonal Efficacy (CSIE-32) | Change from baseline at 20 weeks
  Change in Circumplex Scales of Interpersonal Efficacy: 32-items; scale 0-10; Higher score indicate confidence that one can engage in variety of interpersonal behaviours.
Total cost of costs of rTMS and tDCS administration | Through study completion, an average of 20 weeks
  Total cost of costs of rTMS and tDCS administration
Duration of inpatient hospital stay as recorded by clinical staff | Through study completion, an average of 20 weeks
  Duration of inpatient hospital stay as recorded by clinical staff
Number of re-admissions as reported by clinical staff. | From date of randomization until the date of study completion, assessed up to 20 weeks.
  Number of re-admissions as reported by clinical staff
Number of psychology sessions | Through study completion, an average of 20 weeks
  Number of psychology sessions
Cost of psychology sessions | Through study completion, an average of 20 weeks
  Cost of psychology sessions in $ AUD

CONTACTS AND LOCATIONS:
Overall Officials: Sloane Madden, Assoc. Prof., Principal Investigator — University of Sydney, Ramsay Health Care
Locations (1):
- Northside Clinic, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data though with ethics approval and data transfer agreements required

REFERENCES:
- [Background] Aardoom JJ, Dingemans AE, Slof Op't Landt MC, Van Furth EF. Norms and discriminative validity of the Eating Disorder Examination Questionnaire (EDE-Q). Eat Behav. 2012 Dec;13(4):305-9. doi: 10.1016/j.eatbeh.2012.09.002. Epub 2012 Sep 19. PMID 23121779
- [Background] First MB. Diagnostic and statistical manual of mental disorders, 5th edition, and clinical utility. J Nerv Ment Dis. 2013 Sep;201(9):727-9. doi: 10.1097/NMD.0b013e3182a2168a. No abstract available. PMID 23995026
- [Background] Alonzo A, Fong J, Ball N, Martin D, Chand N, Loo C. Pilot trial of home-administered transcranial direct current stimulation for the treatment of depression. J Affect Disord. 2019 Jun 1;252:475-483. doi: 10.1016/j.jad.2019.04.041. Epub 2019 Apr 10. PMID 31005790
- [Background] Arcelus J, Mitchell AJ, Wales J, Nielsen S. Mortality rates in patients with anorexia nervosa and other eating disorders. A meta-analysis of 36 studies. Arch Gen Psychiatry. 2011 Jul;68(7):724-31. doi: 10.1001/archgenpsychiatry.2011.74. PMID 21727255
- [Background] Berryhill ME, Martin D. Cognitive Effects of Transcranial Direct Current Stimulation in Healthy and Clinical Populations: An Overview. J ECT. 2018 Sep;34(3):e25-e35. doi: 10.1097/YCT.0000000000000534. PMID 30095685
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Couturier J, Lock J. What is remission in adolescent anorexia nervosa? A review of various conceptualizations and quantitative analysis. Int J Eat Disord. 2006 Apr;39(3):175-83. doi: 10.1002/eat.20224. PMID 16485268
- [Background] Dalton B, Bartholdy S, McClelland J, Kekic M, Rennalls SJ, Werthmann J, Carter B, O'Daly OG, Campbell IC, David AS, Glennon D, Kern N, Schmidt U. Randomised controlled feasibility trial of real versus sham repetitive transcranial magnetic stimulation treatment in adults with severe and enduring anorexia nervosa: the TIARA study. BMJ Open. 2018 Jul 16;8(7):e021531. doi: 10.1136/bmjopen-2018-021531. PMID 30012789
- [Background] Dedoncker J, Brunoni AR, Baeken C, Vanderhasselt MA. A Systematic Review and Meta-Analysis of the Effects of Transcranial Direct Current Stimulation (tDCS) Over the Dorsolateral Prefrontal Cortex in Healthy and Neuropsychiatric Samples: Influence of Stimulation Parameters. Brain Stimul. 2016 Jul-Aug;9(4):501-17. doi: 10.1016/j.brs.2016.04.006. Epub 2016 Apr 12. PMID 27160468
- [Background] Fairburn, G.G. Cognitive Behavior Therapy and Eating Disorders. Guilford Press, New York, 2008.
- [Background] Garber AK, Sawyer SM, Golden NH, Guarda AS, Katzman DK, Kohn MR, Le Grange D, Madden S, Whitelaw M, Redgrave GW. A systematic review of approaches to refeeding in patients with anorexia nervosa. Int J Eat Disord. 2016 Mar;49(3):293-310. doi: 10.1002/eat.22482. Epub 2015 Dec 12. PMID 26661289
- [Background] Hatch A, Madden S, Kohn M, Clarke S, Touyz S, Williams LM. Anorexia nervosa: towards an integrative neuroscience model. Eur Eat Disord Rev. 2010 May;18(3):165-79. doi: 10.1002/erv.974. PMID 20443202
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Katzman DK. Medical complications in adolescents with anorexia nervosa: a review of the literature. Int J Eat Disord. 2005;37 Suppl:S52-9; discussion S87-9. doi: 10.1002/eat.20118. PMID 15852321
- [Background] Khedr EM, Elfetoh NA, Ali AM, Noamany M. Anodal transcranial direct current stimulation over the dorsolateral prefrontal cortex improves anorexia nervosa: A pilot study. Restor Neurol Neurosci. 2014;32(6):789-97. doi: 10.3233/RNN-140392. PMID 25189181
- [Background] Knyahnytska YO, Blumberger DM, Daskalakis ZJ, Zomorrodi R, Kaplan AS. Insula H-coil deep transcranial magnetic stimulation in severe and enduring anorexia nervosa (SE-AN): a pilot study. Neuropsychiatr Dis Treat. 2019 Aug 6;15:2247-2256. doi: 10.2147/NDT.S207630. eCollection 2019. PMID 31496707
- [Background] Lewinsohn PM, Striegel-Moore RH, Seeley JR. Epidemiology and natural course of eating disorders in young women from adolescence to young adulthood. J Am Acad Child Adolesc Psychiatry. 2000 Oct;39(10):1284-92. doi: 10.1097/00004583-200010000-00016. PMID 11026183
- [Background] Liu A, Voroslakos M, Kronberg G, Henin S, Krause MR, Huang Y, Opitz A, Mehta A, Pack CC, Krekelberg B, Berenyi A, Parra LC, Melloni L, Devinsky O, Buzsaki G. Immediate neurophysiological effects of transcranial electrical stimulation. Nat Commun. 2018 Nov 30;9(1):5092. doi: 10.1038/s41467-018-07233-7. PMID 30504921
- [Background] Loo CK, Martin DM, Alonzo A, Gandevia S, Mitchell PB, Sachdev P. Avoiding skin burns with transcranial direct current stimulation: preliminary considerations. Int J Neuropsychopharmacol. 2011 Apr;14(3):425-6. doi: 10.1017/S1461145710001197. Epub 2010 Oct 6. No abstract available. PMID 20923600
- [Background] Lovibond, S.H. & Lovibond, P.F. (1995). Manual for the Depression Anxiety Stress Scales. (2nd. Ed.) Sydney: Psychology Foundation.
- [Background] Madden, S. (2015). Biopsychiatric theories of eating disorders. In The Wiley Handbook of Eating Disorders. Assessment, Prevention, Treatment, Policy, and Future Directions, Eds. Smolak, L., and Levine, M.P.
- [Background] Martin DM, McClintock SM, Forster JJ, Lo TY, Loo CK. Cognitive enhancing effects of rTMS administered to the prefrontal cortex in patients with depression: A systematic review and meta-analysis of individual task effects. Depress Anxiety. 2017 Nov;34(11):1029-1039. doi: 10.1002/da.22658. Epub 2017 May 24. PMID 28543994
- [Background] McClelland J, Kekic M, Campbell IC, Schmidt U. Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment in Enduring Anorexia Nervosa: A Case Series. Eur Eat Disord Rev. 2016 Mar;24(2):157-63. doi: 10.1002/erv.2414. Epub 2015 Nov 4. PMID 26537308
- [Background] McClintock SM, Reti IM, Carpenter LL, McDonald WM, Dubin M, Taylor SF, Cook IA, O'Reardon J, Husain MM, Wall C, Krystal AD, Sampson SM, Morales O, Nelson BG, Latoussakis V, George MS, Lisanby SH; National Network of Depression Centers rTMS Task Group; American Psychiatric Association Council on Research Task Force on Novel Biomarkers and Treatments. Consensus Recommendations for the Clinical Application of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Depression. J Clin Psychiatry. 2018 Jan/Feb;79(1):16cs10905. doi: 10.4088/JCP.16cs10905. PMID 28541649
- [Background] Moffa AH, Martin D, Alonzo A, Bennabi D, Blumberger DM, Bensenor IM, Daskalakis Z, Fregni F, Haffen E, Lisanby SH, Padberg F, Palm U, Razza LB, Sampaio-Jr B, Loo C, Brunoni AR. Efficacy and acceptability of transcranial direct current stimulation (tDCS) for major depressive disorder: An individual patient data meta-analysis. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Apr 20;99:109836. doi: 10.1016/j.pnpbp.2019.109836. Epub 2019 Dec 16. PMID 31837388
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Murray SB, Loeb KL, Le Grange D. Treatment outcome reporting in anorexia nervosa: time for a paradigm shift? J Eat Disord. 2018 May 7;6:10. doi: 10.1186/s40337-018-0195-1. eCollection 2018. No abstract available. PMID 29760916
- [Background] Mutz J, Vipulananthan V, Carter B, Hurlemann R, Fu CHY, Young AH. Comparative efficacy and acceptability of non-surgical brain stimulation for the acute treatment of major depressive episodes in adults: systematic review and network meta-analysis. BMJ. 2019 Mar 27;364:l1079. doi: 10.1136/bmj.l1079. PMID 30917990
- [Background] Patel R, Silla F, Pierce S, Theule J, Girard TA. Cognitive functioning before and after repetitive transcranial magnetic stimulation (rTMS): A quantitative meta-analysis in healthy adults. Neuropsychologia. 2020 Apr;141:107395. doi: 10.1016/j.neuropsychologia.2020.107395. Epub 2020 Mar 4. PMID 32142730
- [Background] Reitan, R. (1979). Trail Making Test. Reitan Neuropsychological Laboratory.
- [Background] Rose JS, Vaewsorn A, Rosselli-Navarra F, Wilson GT, Weissman RS. Test-retest reliability of the eating disorder examination-questionnaire (EDE-Q) in a college sample. J Eat Disord. 2013 Nov 20;1:42. doi: 10.1186/2050-2974-1-42. eCollection 2013. PMID 24999420
- [Background] Smith KE, Mason TB, Johnson JS, Lavender JM, Wonderlich SA. A systematic review of reviews of neurocognitive functioning in eating disorders: The state-of-the-literature and future directions. Int J Eat Disord. 2018 Aug;51(8):798-821. doi: 10.1002/eat.22929. Epub 2018 Aug 13. PMID 30102781
- [Background] Steinhausen HC. The outcome of anorexia nervosa in the 20th century. Am J Psychiatry. 2002 Aug;159(8):1284-93. doi: 10.1176/appi.ajp.159.8.1284. PMID 12153817
- [Background] Strumila R, Thiebaut S, Jaussent I, Seneque M, Attal J, Courtet P, Guillaume S. Safety and efficacy of transcranial direct current stimulation (tDCS) in the treatment of Anorexia Nervosa. The open-label STAR study. Brain Stimul. 2019 Sep-Oct;12(5):1325-1327. doi: 10.1016/j.brs.2019.06.017. Epub 2019 Jun 19. No abstract available. PMID 31239105
- [Background] Wade TD, Bergin JL, Tiggemann M, Bulik CM, Fairburn CG. Prevalence and long-term course of lifetime eating disorders in an adult Australian twin cohort. Aust N Z J Psychiatry. 2006 Feb;40(2):121-8. doi: 10.1080/j.1440-1614.2006.01758.x. PMID 16476129
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Westwood H, Stahl D, Mandy W, Tchanturia K. The set-shifting profiles of anorexia nervosa and autism spectrum disorder using the Wisconsin Card Sorting Test: a systematic review and meta-analysis. Psychol Med. 2016 Jul;46(9):1809-27. doi: 10.1017/S0033291716000581. Epub 2016 Apr 25. PMID 27109830
- [Background] Wu M, Giel KE, Skunde M, Schag K, Rudofsky G, de Zwaan M, Zipfel S, Herzog W, Friederich HC. Inhibitory control and decision making under risk in bulimia nervosa and binge-eating disorder. Int J Eat Disord. 2013 Nov;46(7):721-8. doi: 10.1002/eat.22143. Epub 2013 Jun 3. PMID 23729277
- [Derived] Harvey AJ, Madden S, Rodgers A, Bull M, Chatterton ML, Hadzi-Pavlovic D, Loo CK, Martin DM. Randomised controlled trial of neurostimulation for symptoms of anorexia nervosa (TRENA study): study protocol. J Eat Disord. 2023 Dec 8;11(1):218. doi: 10.1186/s40337-023-00940-7. PMID 38066658